CLINICAL TRIAL: NCT02593357
Title: Assessment of a Peripheral Endothelial Dysfunction in COPD (Chronic Obstructive Pulmonary Disease)
Brief Title: Peripheral Endothelial Function in COPD Patients
Acronym: endothBPCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012/55
Record Dates: First submitted 2015-10-16; First posted 2015-11-02 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: endothelial function; COPD; pulmonary function
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COPD patients (Experimental): measure of endothelial function with EndoPAT® in COPD patients
  Interventions: Device: COPD patients

INTERVENTIONS:
Device: COPD patients — measure of peripheral endothelial function by the reactive hyperemia-peripheral artery tone index with a specific device (EndoPAT®)

SUMMARY:
The aim of the study is to assess the peripheral endothelial function in adult COPD (chronic obstructive pulmonary disease) patients and the relationship between the peripheral endothelial function and the pulmonary function.

DETAILED DESCRIPTION:
The primary criteria is the peripheral endothelial function that will be assessed by the measure of flow-mediated dilation (reactive hyperemia-peripheral artery tone index). The pulmonary function will be assessed by the measures of the FEV1 (forced expiratory volume in one second), the forced vital capacity (FVC) and the expiratory flow between 25% and 75% (FEF25-75%). The relationship between these parameters of the pulmonary function and the peripheral endothelial function will be analyzed. In addition, a relationship between peripheral endothelial function and the severity of COPD (classification according to GOLD (Global Initiative for Chronic Obstructive Lung Disease) 2010 and GOLD 2011 and the COPD assessment test, the cardiovascular risk factors (SCORE INdex) and the smoker status will be also assessed.

ELIGIBILITY:
Inclusion Criteria:

* COPD : FEV1/FVC < 70%
* Smokers or ex-smokers ( ≥ 10 pack-years)
* No COPD exacerbation in the last three months
* No history of asthma and no respiratory allergy

Exclusion Criteria:

* Pregnant or nursing women
* Treatment with pulmonary vasodilators
* Patients with a significant acute disease. A significant disease is defined as a disease which, in the opinion of the investigator, may influence the results of the trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2012-12-17 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-08-17 (Actual)

PRIMARY OUTCOMES:
measure of reactive hyperemia-peripheral artery tone index | Day 1
  measure of reactive hyperemia-peripheral artery tone index

SECONDARY OUTCOMES:
measure of Forced expiratory flow in one second | day 1
  measure of Forced expiratory flow in one second
measure of forced vital capacity | day 1
  measure of forced vital capacity
measure of expiratory flow between 25% and 75% (FEF25-75%). | day 1
  measure of expiratory flow between 25% and 75% (FEF25-75%).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Saint-Antoine, Paris
  - Hôpital Foch, Suresnes

REFERENCES:
- [Background] Furchgott RF, Zawadzki JV. The obligatory role of endothelial cells in the relaxation of arterial smooth muscle by acetylcholine. Nature. 1980 Nov 27;288(5789):373-6. doi: 10.1038/288373a0. PMID 6253831
- [Background] Lockette W, Otsuka Y, Carretero O. The loss of endothelium-dependent vascular relaxation in hypertension. Hypertension. 1986 Jun;8(6 Pt 2):II61-6. doi: 10.1161/01.hyp.8.6_pt_2.ii61. PMID 3087875
- [Background] Ibengwe JK, Suzuki H. Changes in mechanical responses of vascular smooth muscles to acetylcholine, noradrenaline and high-potassium solution in hypercholesterolemic rabbits. Br J Pharmacol. 1986 Feb;87(2):395-402. doi: 10.1111/j.1476-5381.1986.tb10829.x. PMID 3955307
- [Background] Santos S, Peinado VI, Ramirez J, Melgosa T, Roca J, Rodriguez-Roisin R, Barbera JA. Characterization of pulmonary vascular remodelling in smokers and patients with mild COPD. Eur Respir J. 2002 Apr;19(4):632-8. doi: 10.1183/09031936.02.00245902. PMID 11998991
- [Background] Henno P, Boitiaux JF, Douvry B, Cazes A, Levy M, Devillier P, Delclaux C, Israel-Biet D. Tobacco-associated pulmonary vascular dysfunction in smokers: role of the ET-1 pathway. Am J Physiol Lung Cell Mol Physiol. 2011 Jun;300(6):L831-9. doi: 10.1152/ajplung.00251.2010. Epub 2011 Mar 4. PMID 21378026
- [Background] Duong-Quy S, Dao P, Hua-Huy T, Guilluy C, Pacaud P, Dinh-Xuan AT. Increased Rho-kinase expression and activity and pulmonary endothelial dysfunction in smokers with normal lung function. Eur Respir J. 2011 Feb;37(2):349-55. doi: 10.1183/09031936.00056610. Epub 2010 Jun 7. PMID 20530044
- [Background] Celermajer DS, Sorensen KE, Georgakopoulos D, Bull C, Thomas O, Robinson J, Deanfield JE. Cigarette smoking is associated with dose-related and potentially reversible impairment of endothelium-dependent dilation in healthy young adults. Circulation. 1993 Nov;88(5 Pt 1):2149-55. doi: 10.1161/01.cir.88.5.2149. PMID 8222109
- [Background] Zeiher AM, Schachinger V, Minners J. Long-term cigarette smoking impairs endothelium-dependent coronary arterial vasodilator function. Circulation. 1995 Sep 1;92(5):1094-100. doi: 10.1161/01.cir.92.5.1094. PMID 7648652
- [Background] Fratta Pasini A, Albiero A, Stranieri C, Cominacini M, Pasini A, Mozzini C, Vallerio P, Cominacini L, Garbin U. Serum oxidative stress-induced repression of Nrf2 and GSH depletion: a mechanism potentially involved in endothelial dysfunction of young smokers. PLoS One. 2012;7(1):e30291. doi: 10.1371/journal.pone.0030291. Epub 2012 Jan 17. PMID 22272327
- [Background] Nana-Sinkam SP, Lee JD, Sotto-Santiago S, Stearman RS, Keith RL, Choudhury Q, Cool C, Parr J, Moore MD, Bull TM, Voelkel NF, Geraci MW. Prostacyclin prevents pulmonary endothelial cell apoptosis induced by cigarette smoke. Am J Respir Crit Care Med. 2007 Apr 1;175(7):676-85. doi: 10.1164/rccm.200605-724OC. Epub 2007 Jan 25. PMID 17255567
- [Background] Hurlimann D, Forster A, Noll G, Enseleit F, Chenevard R, Distler O, Bechir M, Spieker LE, Neidhart M, Michel BA, Gay RE, Luscher TF, Gay S, Ruschitzka F. Anti-tumor necrosis factor-alpha treatment improves endothelial function in patients with rheumatoid arthritis. Circulation. 2002 Oct 22;106(17):2184-7. doi: 10.1161/01.cir.0000037521.71373.44. PMID 12390945
- [Background] Peinado VI, Barbera JA, Ramirez J, Gomez FP, Roca J, Jover L, Gimferrer JM, Rodriguez-Roisin R. Endothelial dysfunction in pulmonary arteries of patients with mild COPD. Am J Physiol. 1998 Jun;274(6):L908-13. doi: 10.1152/ajplung.1998.274.6.L908. PMID 9609729
- [Background] Hughes R, Tong J, Oates C, Lordan J, Corris PA. Evidence for systemic endothelial dysfunction in patients and first-order relatives with pulmonary arterial hypertension. Chest. 2005 Dec;128(6 Suppl):617S. doi: 10.1378/chest.128.6_suppl.617S. No abstract available. PMID 16373872
- [Background] Wolff B, Lodziewski S, Bollmann T, Opitz CF, Ewert R. Impaired peripheral endothelial function in severe idiopathic pulmonary hypertension correlates with the pulmonary vascular response to inhaled iloprost. Am Heart J. 2007 Jun;153(6):1088.e1-7. doi: 10.1016/j.ahj.2007.03.005. PMID 17540215
- [Background] Peled N, Bendayan D, Shitrit D, Fox B, Yehoshua L, Kramer MR. Peripheral endothelial dysfunction in patients with pulmonary arterial hypertension. Respir Med. 2008 Dec;102(12):1791-6. doi: 10.1016/j.rmed.2008.06.014. Epub 2008 Aug 3. PMID 18678478
- [Background] Dorfmuller P, Perros F, Balabanian K, Humbert M. Inflammation in pulmonary arterial hypertension. Eur Respir J. 2003 Aug;22(2):358-63. doi: 10.1183/09031936.03.00038903. PMID 12952274
- [Background] Friedman R, Mears JG, Barst RJ. Continuous infusion of prostacyclin normalizes plasma markers of endothelial cell injury and platelet aggregation in primary pulmonary hypertension. Circulation. 1997 Nov 4;96(9):2782-4. doi: 10.1161/01.cir.96.9.2782. PMID 9386137
- [Background] Christman BW, McPherson CD, Newman JH, King GA, Bernard GR, Groves BM, Loyd JE. An imbalance between the excretion of thromboxane and prostacyclin metabolites in pulmonary hypertension. N Engl J Med. 1992 Jul 9;327(2):70-5. doi: 10.1056/NEJM199207093270202. PMID 1603138
- [Background] Xu W, Kaneko FT, Zheng S, Comhair SA, Janocha AJ, Goggans T, Thunnissen FB, Farver C, Hazen SL, Jennings C, Dweik RA, Arroliga AC, Erzurum SC. Increased arginase II and decreased NO synthesis in endothelial cells of patients with pulmonary arterial hypertension. FASEB J. 2004 Nov;18(14):1746-8. doi: 10.1096/fj.04-2317fje. Epub 2004 Sep 13. PMID 15364894
- [Background] Celli BR, MacNee W; ATS/ERS Task Force. Standards for the diagnosis and treatment of patients with COPD: a summary of the ATS/ERS position paper. Eur Respir J. 2004 Jun;23(6):932-46. doi: 10.1183/09031936.04.00014304. No abstract available. PMID 15219010
- [Background] Anthonisen NR, Connett JE, Enright PL, Manfreda J; Lung Health Study Research Group. Hospitalizations and mortality in the Lung Health Study. Am J Respir Crit Care Med. 2002 Aug 1;166(3):333-9. doi: 10.1164/rccm.2110093. PMID 12153966
- [Background] Sin DD, Wu L, Man SF. The relationship between reduced lung function and cardiovascular mortality: a population-based study and a systematic review of the literature. Chest. 2005 Jun;127(6):1952-9. doi: 10.1378/chest.127.6.1952. PMID 15947307
- [Background] Tockman MS, Pearson JD, Fleg JL, Metter EJ, Kao SY, Rampal KG, Cruise LJ, Fozard JL. Rapid decline in FEV1. A new risk factor for coronary heart disease mortality. Am J Respir Crit Care Med. 1995 Feb;151(2 Pt 1):390-8. doi: 10.1164/ajrccm.151.2.7842197.
- [Background] Johnston AK, Mannino DM, Hagan GW, Davis KJ, Kiri VA. Relationship between lung function impairment and incidence or recurrence of cardiovascular events in a middle-aged cohort. Thorax. 2008 Jul;63(7):599-605. doi: 10.1136/thx.2007.088112. Epub 2008 Feb 1. PMID 18245145
- [Background] Gan WQ, Man SF, Senthilselvan A, Sin DD. Association between chronic obstructive pulmonary disease and systemic inflammation: a systematic review and a meta-analysis. Thorax. 2004 Jul;59(7):574-80. doi: 10.1136/thx.2003.019588. PMID 15223864
- [Background] Sin DD, Man SF. Why are patients with chronic obstructive pulmonary disease at increased risk of cardiovascular diseases? The potential role of systemic inflammation in chronic obstructive pulmonary disease. Circulation. 2003 Mar 25;107(11):1514-9. doi: 10.1161/01.cir.0000056767.69054.b3. PMID 12654609
- [Background] Pinto-Plata VM, Mullerova H, Toso JF, Feudjo-Tepie M, Soriano JB, Vessey RS, Celli BR. C-reactive protein in patients with COPD, control smokers and non-smokers. Thorax. 2006 Jan;61(1):23-8. doi: 10.1136/thx.2005.042200. Epub 2005 Sep 2. PMID 16143583
- [Background] Macnee W, Maclay J, McAllister D. Cardiovascular injury and repair in chronic obstructive pulmonary disease. Proc Am Thorac Soc. 2008 Dec 1;5(8):824-33. doi: 10.1513/pats.200807-071TH. PMID 19017737
- [Background] Zureik M, Benetos A, Neukirch C, Courbon D, Bean K, Thomas F, Ducimetiere P. Reduced pulmonary function is associated with central arterial stiffness in men. Am J Respir Crit Care Med. 2001 Dec 15;164(12):2181-5. doi: 10.1164/ajrccm.164.12.2107137. PMID 11751184
- [Background] Zureik M, Kauffmann F, Touboul PJ, Courbon D, Ducimetiere P. Association between peak expiratory flow and the development of carotid atherosclerotic plaques. Arch Intern Med. 2001 Jul 9;161(13):1669-76. doi: 10.1001/archinte.161.13.1669. PMID 11434800
- [Background] Taneda K, Namekata T, Hughes D, Suzuki K, Knopp R, Ozasa K. Association of lung function with atherosclerotic risk factors among Japanese Americans: Seattle Nikkei Health Study. Clin Exp Pharmacol Physiol. 2004 Dec;31 Suppl 2:S31-4. doi: 10.1111/j.1440-1681.2004.04116.x. PMID 15649282
- [Background] Maclay JD, McAllister DA, Mills NL, Paterson FP, Ludlam CA, Drost EM, Newby DE, Macnee W. Vascular dysfunction in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Sep 15;180(6):513-20. doi: 10.1164/rccm.200903-0414OC. Epub 2009 Jun 19. PMID 19542477
- [Background] Janner JH, McAllister DA, Godtfredsen NS, Prescott E, Vestbo J. Is chronic obstructive pulmonary disease associated with increased arterial stiffness? Respir Med. 2012 Mar;106(3):397-405. doi: 10.1016/j.rmed.2011.08.016. Epub 2011 Dec 3. PMID 22136986
- [Background] Barr RG, Mesia-Vela S, Austin JH, Basner RC, Keller BM, Reeves AP, Shimbo D, Stevenson L. Impaired flow-mediated dilation is associated with low pulmonary function and emphysema in ex-smokers: the Emphysema and Cancer Action Project (EMCAP) Study. Am J Respir Crit Care Med. 2007 Dec 15;176(12):1200-7. doi: 10.1164/rccm.200707-980OC. Epub 2007 Aug 29. PMID 17761614
- [Background] Heitzer T, Schlinzig T, Krohn K, Meinertz T, Munzel T. Endothelial dysfunction, oxidative stress, and risk of cardiovascular events in patients with coronary artery disease. Circulation. 2001 Nov 27;104(22):2673-8. doi: 10.1161/hc4601.099485. PMID 11723017
- [Background] Suwaidi JA, Hamasaki S, Higano ST, Nishimura RA, Holmes DR Jr, Lerman A. Long-term follow-up of patients with mild coronary artery disease and endothelial dysfunction. Circulation. 2000 Mar 7;101(9):948-54. doi: 10.1161/01.cir.101.9.948. PMID 10704159
- [Background] Celermajer DS, Sorensen KE, Gooch VM, Spiegelhalter DJ, Miller OI, Sullivan ID, Lloyd JK, Deanfield JE. Non-invasive detection of endothelial dysfunction in children and adults at risk of atherosclerosis. Lancet. 1992 Nov 7;340(8828):1111-5. doi: 10.1016/0140-6736(92)93147-f. PMID 1359209
- [Background] Asmar R, Benetos A, Topouchian J, Laurent P, Pannier B, Brisac AM, Target R, Levy BI. Assessment of arterial distensibility by automatic pulse wave velocity measurement. Validation and clinical application studies. Hypertension. 1995 Sep;26(3):485-90. doi: 10.1161/01.hyp.26.3.485. PMID 7649586
- [Background] Hayward CS, Kraidly M, Webb CM, Collins P. Assessment of endothelial function using peripheral waveform analysis: a clinical application. J Am Coll Cardiol. 2002 Aug 7;40(3):521-8. doi: 10.1016/s0735-1097(02)01991-5. PMID 12142121
- [Background] Hamburg NM, Keyes MJ, Larson MG, Vasan RS, Schnabel R, Pryde MM, Mitchell GF, Sheffy J, Vita JA, Benjamin EJ. Cross-sectional relations of digital vascular function to cardiovascular risk factors in the Framingham Heart Study. Circulation. 2008 May 13;117(19):2467-74. doi: 10.1161/CIRCULATIONAHA.107.748574. Epub 2008 May 5. PMID 18458169
- [Background] Flammer AJ, Anderson T, Celermajer DS, Creager MA, Deanfield J, Ganz P, Hamburg NM, Luscher TF, Shechter M, Taddei S, Vita JA, Lerman A. The assessment of endothelial function: from research into clinical practice. Circulation. 2012 Aug 7;126(6):753-67. doi: 10.1161/CIRCULATIONAHA.112.093245. PMID 22869857
- [Background] Selamet Tierney ES, Newburger JW, Gauvreau K, Geva J, Coogan E, Colan SD, de Ferranti SD. Endothelial pulse amplitude testing: feasibility and reproducibility in adolescents. J Pediatr. 2009 Jun;154(6):901-5. doi: 10.1016/j.jpeds.2008.12.028. Epub 2009 Feb 12. PMID 19217124
- [Background] Dhindsa M, Sommerlad SM, DeVan AE, Barnes JN, Sugawara J, Ley O, Tanaka H. Interrelationships among noninvasive measures of postischemic macro- and microvascular reactivity. J Appl Physiol (1985). 2008 Aug;105(2):427-32. doi: 10.1152/japplphysiol.90431.2008. Epub 2008 May 15. PMID 18483158
- [Background] Kuvin JT, Patel AR, Sliney KA, Pandian NG, Sheffy J, Schnall RP, Karas RH, Udelson JE. Assessment of peripheral vascular endothelial function with finger arterial pulse wave amplitude. Am Heart J. 2003 Jul;146(1):168-74. doi: 10.1016/S0002-8703(03)00094-2. PMID 12851627
- [Background] Nohria A, Gerhard-Herman M, Creager MA, Hurley S, Mitra D, Ganz P. Role of nitric oxide in the regulation of digital pulse volume amplitude in humans. J Appl Physiol (1985). 2006 Aug;101(2):545-8. doi: 10.1152/japplphysiol.01285.2005. Epub 2006 Apr 13. PMID 16614356
- [Background] Bonetti PO, Pumper GM, Higano ST, Holmes DR Jr, Kuvin JT, Lerman A. Noninvasive identification of patients with early coronary atherosclerosis by assessment of digital reactive hyperemia. J Am Coll Cardiol. 2004 Dec 7;44(11):2137-41. doi: 10.1016/j.jacc.2004.08.062. PMID 15582310
- [Background] Mahmud FH, Van Uum S, Kanji N, Thiessen-Philbrook H, Clarson CL. Impaired endothelial function in adolescents with type 1 diabetes mellitus. J Pediatr. 2008 Apr;152(4):557-62. doi: 10.1016/j.jpeds.2007.08.044. Epub 2007 Nov 5. PMID 18346515
- [Background] Lowenstein L, Damti A, Pillar G, Shott S, Blumenfeld Z. Evaluation of endothelial function in women with polycystic ovary syndrome. Eur J Obstet Gynecol Reprod Biol. 2007 Oct;134(2):208-12. doi: 10.1016/j.ejogrb.2007.02.011. Epub 2007 Mar 19. PMID 17374431
- [Background] Roifman I, Sun YC, Fedwick JP, Panaccione R, Buret AG, Liu H, Rostom A, Anderson TJ, Beck PL. Evidence of endothelial dysfunction in patients with inflammatory bowel disease. Clin Gastroenterol Hepatol. 2009 Feb;7(2):175-82. doi: 10.1016/j.cgh.2008.10.021. Epub 2008 Oct 30. PMID 19121648
- [Background] Itzhaki S, Lavie L, Pillar G, Tal G, Lavie P. Endothelial dysfunction in obstructive sleep apnea measured by peripheral arterial tone response in the finger to reactive hyperemia. Sleep. 2005 May;28(5):594-600. doi: 10.1093/sleep/28.5.594. PMID 16171272